CLINICAL TRIAL: NCT00728715
Title: Clinical Efficacy and Safety of Budesonide and Formoterol in the Management of Non-Cystic Fibrosis Bronchiectasis
Brief Title: Efficacy of Budesonide-Formoterol in Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General de Requena (Other)
Collaborators: Esteve (Other)
Responsible Party: Dr Miguel Angel Martínez-Garcia, Hospital General de Requena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGR-0000013
Record Dates: First submitted 2008-07-31; First posted 2008-08-06 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 2008-07

CONDITIONS: Bronchiectasis
Keywords: Budesonide; Formoterol; Non cystic fibrosis bronchiectasis
MeSH Terms: conditions — Bronchiectasis | interventions — Formoterol Fumarate; Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Medium Dose of budesonide-formoterol
  Interventions: Drug: budesonide-formoterol single inhaler; Drug: High dose of budesonide; Drug: A
- B (Active Comparator): High dose of inhaled budesonide (1600 mcg/day)
  Interventions: Drug: budesonide-formoterol single inhaler; Drug: High dose of budesonide; Drug: B

INTERVENTIONS:
Drug: budesonide-formoterol single inhaler — High dose budesonide:Budesonide (Pulmocort turbuhaler) 400 mcg (2 inhalations bid) Medium dose budesonide plus formoterol (Rilast turbuhaler) 4,5 mcg of formoterol plus 400 mcg of budesonide: 2 inhalations bid
  Other Names: B. High-dose budesonide arm; A. Medium dose of budesonide plus formoterol
Drug: High dose of budesonide — 1600 mcg/d of budesonide
Drug: A — medium dose of budesonide-formoterol
  Arms: A
Drug: B — High Dose Inhaled Budesonide
  Arms: B

SUMMARY:
Some studies have concluded that high-dose inhaled steroids (IS) are effective in the clinical control of patients with bronchiectasis, however the high doses needed provokes some adverse effects and lower doses are not effective. Combined treatment with budesonide and formoterol have demostrated to be effective in patients with asthma and COPD achieving the reduction of steroid dose thanks to the adition of a long-acting beta 2 agonists. There are no studies in the literature analysing the effect of combined treatment in patients with bronchiectasis. The objective of this study is to compare the efficacy and safety of formoterol-medium dose of budesonide in a single inhaler versus high-dose of budesonide in the clinical control of patientes with non-cystic fibrosis bronchiectasis.

Study Design:

Randomized (3 months) parallel groups study.

Patients:

Patients with bronchiectasis diagnosed by high-resolution CT scan and chronic obstructive airway obstruction.

Exclusion:

Asthma and current or past smokers.

Methods:

Run in period in all patients with high dose of budesonide (1600 mcg/day) for 3 months. After that, randomization into two groups: 1. The same treatment (1600 mcg/day of budesonide) or combined treatment with lower dose of budesonide (18 mcg/day of formoterol and 800 mcg of budesonide) in a single turbuhaler inhaler during 3 months.

Studied variables:

Clinical, functional, quality of life, microbiological and number of side effects.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old patients diagnosed of non-cystic fibrosis bronchiectasis
* More than 1 pulmonary lobe affected
* Chronic obstructive airflow obstruction
* Stable phase of the disease

Exclusion Criteria:

* Asthma, COPD or current/past smnokers
* No consent
* Known intolerance to budesonide or formoterol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-01; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Health related quality of life (measured by St Gorge Respiratory Questionnaire) | at 3 and 6 months

SECONDARY OUTCOMES:
Forced spirometry; microbiological data, clinical data (dyspnea, cough, wheezes) and side effects | at 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General de Requena, Valencia, Valencia, Spain

REFERENCES:
- [Derived] Martinez-Garcia MA, Soler-Cataluna JJ, Catalan-Serra P, Roman-Sanchez P, Tordera MP. Clinical efficacy and safety of budesonide-formoterol in non-cystic fibrosis bronchiectasis. Chest. 2012 Feb;141(2):461-468. doi: 10.1378/chest.11-0180. Epub 2011 Jul 21. PMID 21778259